CLINICAL TRIAL: NCT04020354
Title: Functional, Neuroplastic and Biomechanical Changes Induced by Early Hand and Arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE) in Pre-school Children With Uni- and Bilateral Cerebral Palsy
Brief Title: Changes Induced by Early HABIT-ILE in Pre-school Children With Uni- and Bilateral Cerebral Palsy
Acronym: EarlyHABIT-ILE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Université Catholique de Louvain (Other)
Collaborators: University Hospital, Brest (Other); University of Pisa (Other); University Hospital, Angers (Other Government); University of Lausanne Hospitals (Other); University of the Balearic Islands (Other); Fondation Paralysie Cérébrale (Other)
Responsible Party: Principal Investigator, Yannick Bleyenheuft, Professor, Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B403201316810d
Record Dates: First submitted 2018-11-20; First posted 2019-07-16 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Cerebral Palsy
Keywords: motor skill learning; functional changes; neuroplastic changes; biomechanical changes
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HABIT-ILE (Experimental): Early HABIT-ILE (Hand and arm bimanual intensive therapy including lower extremities) will be applied over 2 weeks.
  Interventions: Behavioral: HABIT-ILE
- Usual Care (Active Comparator): A two weeks period of usual customary care
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: HABIT-ILE — Early Hand and arm bimanual intensive therapy including lower extremities
  Arms: HABIT-ILE
Behavioral: Usual Care — Usual customary care
  Arms: Usual Care

SUMMARY:
Studying in two randomized controlled trials (RCT) the changes induced by early HABIT-ILE in functional, neuroplastic and biomechanical assessment in children with unilateral and bilateral CP.

DETAILED DESCRIPTION:
This study aims to evaluate the effect of two weeks of early Hand-arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE) on bimanual performance in pre-school children with unilateral cerebral palsy (CP) and on gross motor function in those with bilateral CP, compared with two weeks of usual motor activity including usual rehabilitation (control group). We will assess further changes in unilateral performance tests, daily life activities questionnaires and executive function tests. Neuroplastic changes will be assessed using brain imaging (magnetic resonance imaging, MRI) and biomechanical changes will be assessed by using optoelectronic motion capture system with electromyography (EMG), to determine the effect of HABIT-ILE on movement pattern and quality.

ELIGIBILITY:
Inclusion Criteria:

* children with unilateral or bilateral cerebral palsy (spastic or dyskinetic)
* age 1 to 4 years inclusive (corrected age if preterm birth)
* ability to follow instructions and complete testing according to the age.

Exclusion Criteria:

* active seizure
* programmed botulinum toxin or orthopedic surgery in the 6 months previous to the intervention, during intervention period or 3months after the intervention time
* severe visual impairments
* severe cognitive impairments
* contraindications to perform MRI assessments (Metal implants, etc.)

Ages: 12 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2018-11-27 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change on Gross Motor Function (GMFM-66) | pre-camp, two weeks post-camp, 3 months follow-up.
  Developed to assess the changes in gross motor function of children with cerebral palsy (scored in percentage), observed over time or after intervention for the second randomized controlled trial (RCT2)
Change on Manual Ability (Assisting Hand Assessment (AHA)) | pre-camp, two weeks post-camp, 3 months follow-up
  Developed to observe the efficacy of the assisting hand use, in children with unilateral cerebral palsy (scored in percentage), during bimanual activities for the first randomized controlled trial (RCT1)

SECONDARY OUTCOMES:
Melbourne 2 Assessment (MA2) | pre-camp, two weeks post-camp, 3 months follow-up
  assess the unilateral performance of the upper extremities, quantifying the dexterity, fluency, accuracy and range of movement during several tasks of reaching and manipulation
Inhibitory control task | pre-camp, two weeks post-camp, 3 months follow-up
  Measures the inhibition of a motor answer. It's assessed by asking the child not to reach for a toy previously showed to play with. The maximum waiting time is 30 seconds.
Working memory task | pre-camp, two weeks post-camp, 3 months follow-up
  Measures the capacity to retain visual information in use, in a short period of time. It's assessed by hiding a toy in front of the child and asking him/her to find it from 4 possibilities.
Visuo-spatial attention assessment | pre-camp, two weeks post-camp, 3 months follow-up
  Through different simple tasks, measures the visual field, the visuo-motor coordination, the orientation of attention in the space and the eye pursuit.
Semmes-Weinstein monofilaments | pre-camp, two weeks post-camp, 3 months follow-up
  Evaluates the pressure threshold or the response to a touching sensation of the filament. It is quantified using a numerical grading ranging from high pression/clear touching sensation to a slight pression/slight touching sensation.
Pressure Threshold | pre-camp, two weeks post-camp, 3 months follow-up
  The superior pressure threshold will be determined at the moment of any visible change in the child's reaction to the pression made by the algometer.
Activlim-CP questionnaire | pre-camp, two weeks post-camp, 3 months follow-up
  This parent's filled questionnaire measures a patient's ability to perform daily activities requiring the use of the upper and/or the lower extremities through 43 items specific to patients with cerebral palsy. It ranges from - 7 to +7 logits (higher score means better performance).
Pediatric Evaluation of Disability Inventory questionnaire (PEDI) | pre-camp, two weeks post-camp, 3 months follow-up
  This parent's filled questionnaire measures the performance of the child in the daily life activities and movement domains, focusing on the capacity of upper extremities and lower extremities during this activities. It ranges from 0 to 100% (higher score means better performance).
Young children's participation and environment measure (YC-PEM) | pre-camp, two weeks post-camp, 3 months follow-up
  Based in different children's activities, this parent's filled questionnaire evaluates the level of participation and the quality of the environment in which these activities take place. For each type of activity, caregivers assess 3 dimensions of the child's participation: frequency (8-point scale; 0-7), level of involvement (5-point scale; 1-5), caregiver's percent desire for change (2-points level (y/n) transformed in percentage; 0-100) and perceived impact of environmental support (3-point scale transformed in percentage; 0-100). A software calculates the total score with a maximum of 212 (higher score means better performance).
Measure of Processes of Care (MPOC-20) | pre-camp, two weeks post-camp, 3 months follow-up
  Assesses the parents' perceptions of the care they and their children receive from children's rehabilitation treatment centres. Using a 8-point response scale, parents answer to 20 questions, indicating to what extent they have experienced the events or the situations described. A score of 7 means that they have experienced this aspect to a very great extent, or most of the time. A score of 1 means that they have not experienced this aspect at all. A score of 0 means that the question does not apply to them.
  There is no total score. However, because the statements are positively worded, higher total scores indicates that needs of the parents are being met to a great extent.
Canadian Occupational Performance Measure (COPM) | pre-camp, two weeks post-camp, 3 months follow-up
  This is an interview-setting designed to capture a patient's self-perception of performance and satisfaction of it in everyday activities, observed over time. During the interview, parents set up 5 activities considered difficult in daily life. These are then assessed, in a 1 to 10 scale, regarding the child's self-perception of performance and satisfaction of it. The total score is the average of the scores for perception and satisfaction separately (score from 1 to 10; higher score means better performance/satisfaction)
3D T1-weighted structural imaging (T1) | pre-camp, 3 months follow-up
  This sequence allows to measure changes in gray matter (cortical thickness)
Changes on the Fractional Anisotropy (Diffusion tensor imaging (DTI)) | pre-camp, 3 months follow-up
  This sequence allows to measure changes in the fractional anisotropy (FA) on the white matter tracts. FA is a scalar value (no unit) between zero and one that describes the degree of anisotropy of white matter water molecules.
Changes on the Mean Diffusivity (Diffusion tensor imaging (DTI)) | pre-camp, 3 months follow-up
  This sequence allows to measure the mean changes in the diffusivity (MD). MD is a scalar value (no unit) between zero and one that describes the degree of molecular diffusion.
Changes on resting state functional connectivity (RS) | pre-camp, 3 months follow-up
  Resting-state functional magnetic resonane imaging (rs-fMRI) evaluates the regional interactions that occur during the resting or task-negative state. The magnitud of the brain activation during rs-fMRI will be assessed
Changes on spatial parameters of the gait (Kinematics assessments) | pre-camp, 3 months follow-up
  Through a 3D motion system, we measure the stride length (meters), step length (meters) and step width (meters).
Changes on temporal parameters of the gait (Cycle time) | pre-camp, 3 months follow-up
  Through a 3D motion system, we measure cycle of gait time (seconds).
Changes on temporal parameters of the gait (Stance time) | pre-camp, 3 months follow-up
  Through a 3D motion system, we measure the stance time (percentage of total gait cycle).
Changes on temporal parameters of the gait (Swing time) | pre-camp, 3 months follow-up
  Through a 3D motion system, we measure the swing time (percentage of total gait cycle).
Changes on temporal parameters of the gait (Stride) | pre-camp, 3 months follow-up
  Through a 3D motion system, we measure the gait cadence (stride per minute).
Changes on temporal parameters of the gait (Velocity) | pre-camp, 3 months follow-up
  Through a 3D motion system, we measure the gait velocity (meter/second)
Changes on temporal parameters of the gait (Acceleration) | pre-camp, 3 months follow-up
  Through a 3D motion system, we measure the gait acceleration (meters/second^2)
Changes on spatial parameters of the upper extremity (Straightness) | pre-camp, 3 months follow-up
  Through a 3D motion system, we measure the straightness (percentage of upper extremity trajectory during a reaching task).
Changes on spatial parameters of the upper extremity (Smoothness) | pre-camp, 3 months follow-up
  Through a 3D motion system, we measure the smoothness (variability of the movement during a reaching task)
Changes on temporal parameters of the upper extremity (Kinematics assessments) | pre-camp, 3 months follow-up
  Through a 3D motion system, we measure the time from onset to end of the task (seconds). the task consist in a reaching task.
Quantification of physical activity | 5 hours during 5 consecutive days
  With a movement sensor on each wrist, the percentage of total time spent in movement (i.e. crawling, walking and running) is measured. Calculated in terms of the changes in the acceleration (m/s^2). These measurements will be performed during therapy in 5 consecutive days for the HABIT-ILE group and during a regular week for the Usual Care group.

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Bleyenheuft, Pr, Principal Investigator — MSL-IN Lab, Institute of Neuroscience, Université catholique de Louvain
Locations (3):
- Institute of Neuroscience, Université catholique de Louvain, Brussels, Belgium
- Fondation ILDYS - Site de Ty Yann, Brest, France
- IRCCS Fondazione Stella Maris, Tirrenia, Tuscany, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Araneda R, Ebner-Karestinos D, Paradis J, Klocker A, Saussez G, Demas J, Bailly R, Bouvier S, Carton de Tournai A, Herman E, Souki A, Le Gal G, Nowak E, Sizonenko SV, Newman CJ, Dinomais M, Riquelme I, Guzzetta A, Brochard S, Bleyenheuft Y. Changes Induced by Early Hand-Arm Bimanual Intensive Therapy Including Lower Extremities in Young Children With Unilateral Cerebral Palsy: A Randomized Clinical Trial. JAMA Pediatr. 2024 Jan 1;178(1):19-28. doi: 10.1001/jamapediatrics.2023.4809. PMID 37930692
- [Derived] Araneda R, Sizonenko SV, Newman CJ, Dinomais M, Le Gal G, Nowak E, Guzzetta A, Riquelme I, Brochard S, Bleyenheuft Y; Early HABIT-ILE group. Functional, neuroplastic and biomechanical changes induced by early Hand-Arm Bimanual Intensive Therapy Including Lower Extremities (e-HABIT-ILE) in pre-school children with unilateral cerebral palsy: study protocol of a randomized control trial. BMC Neurol. 2020 Apr 14;20(1):133. doi: 10.1186/s12883-020-01705-4. PMID 32290815